CLINICAL TRIAL: NCT00008359
Title: A Multicenter, Double-Blind, Randomized, Comparative Study To Evaluate The Safety, Tolerability, And Efficacy Of MK-0991 Versus (Amphotericin B) Liposome For Injection As Empirical Therapy In Patients With Persistent Fever And Neutropenia
Brief Title: Caspofungin Acetate Compared With Amphotericin B Liposomal in Treating Patients With Persistent Fever and Neutropenia Following Cancer Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: 00-085; MSKCC-00085; MERCK-026-01; NCI-G00-1898
Record Dates: First submitted 2001-01-06; First posted 2003-09-04 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Cancer
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; stage IV breast cancer; stage IIIA breast cancer; monoclonal gammopathy of undetermined significance; stage IIIB breast cancer; recurrent adult Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; isolated plasmacytoma of bone; extramedullary plasmacytoma; refractory multiple myeloma; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; disseminated neuroblastoma; recurrent neuroblastoma; recurrent Wilms tumor and other childhood kidney tumors; stage 0 chronic lymphocytic leukemia; Waldenstrom macroglobulinemia; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; small intestine lymphoma; stage III malignant testicular germ cell tumor; recurrent malignant testicular germ cell tumor; unspecified adult solid tumor, protocol specific; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; polycythemia vera; primary myelofibrosis; essential thrombocythemia; fever, sweats, and hot flashes; testicular embryonal carcinoma; testicular choriocarcinoma; testicular teratoma; testicular yolk sac tumor; testicular embryonal carcinoma and teratoma; testicular embryonal carcinoma and teratoma with seminoma; testicular embryonal carcinoma and yolk sac tumor; testicular embryonal carcinoma and yolk sac tumor with seminoma; testicular embryonal carcinoma and seminoma; testicular yolk sac tumor and teratoma; testicular yolk sac tumor and teratoma with seminoma; testicular choriocarcinoma and yolk sac tumor; testicular choriocarcinoma and embryonal carcinoma; testicular choriocarcinoma and teratoma; testicular choriocarcinoma and seminoma; progressive hairy cell leukemia, initial treatment; refractory hairy cell leukemia; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult Burkitt lymphoma; recurrent ovarian germ cell tumor; chronic myelomonocytic leukemia; T-cell large granular lymphocyte leukemia; ovarian yolk sac tumor; ovarian embryonal carcinoma; ovarian polyembryoma; ovarian choriocarcinoma; ovarian immature teratoma; ovarian mature teratoma; ovarian monodermal and highly specialized teratoma; ovarian mixed germ cell tumor; acute undifferentiated leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; high risk metastatic gestational trophoblastic tumor; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; primary central nervous system non-Hodgkin lymphoma; neutropenia; infection; prolymphocytic leukemia; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; primary systemic amyloidosis; intraocular lymphoma; stage I mantle cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Neoplasms; Hodgkin Disease; Breast Neoplasms; Monoclonal Gammopathy of Undetermined Significance; Lymphoma, T-Cell, Cutaneous; Multiple Myeloma; Carcinoma, Ovarian Epithelial; Neuroblastoma; Wilms Tumor; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Testicular Neoplasms; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Polycythemia Vera; Primary Myelofibrosis; Thrombocythemia, Essential; Fever; Hot Flashes; Teratoma, Testicular; Endodermal Sinus Tumor; Teratoma; Seminoma; Carcinoma, Embryonal; Leukemia, Hairy Cell; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Leukemia, Myelomonocytic, Chronic; Leukemia, Large Granular Lymphocytic; Leukemia, Biphenotypic, Acute; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Neutropenia; Infections; Leukemia, Prolymphocytic; Immunoglobulin Light-chain Amyloidosis; Intraocular Lymphoma; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone | interventions — Caspofungin; liposomal amphotericin B

INTERVENTIONS:
Drug: caspofungin acetate
Drug: liposomal amphotericin B

SUMMARY:
RATIONALE: Caspofungin acetate or amphotericin B liposomal may be effective in preventing or controlling fever and neutropenia caused by chemotherapy, bone marrow transplantation, or peripheral stem cell transplantation. It is not yet known whether caspofungin acetate or amphotericin B liposomal is more effective for treating these side effects.

PURPOSE: Randomized phase III trial to compare the effectiveness of caspofungin acetate with that of amphotericin B liposomal in treating patients who have persistent fever and neutropenia after receiving anticancer therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the number of successful treatment outcomes among patients treated with caspofungin acetate vs amphotericin B liposomal for persistent fever and neutropenia following cancer therapy, in terms of survival for 7 days after study drug, resolution of fever, treatment of any baseline fungal infection, absence of breakthrough fungal infection during and for 7 days after study drug, and absence of study drug discontinuation due to toxicity or lack of efficacy.
* Compare the incidence of nephrotoxicity in patients treated with these regimens.
* Compare the incidence of infusion-related adverse events within 1 hour of the infusion in patients treated with these regimens.
* Compare the incidence of treatment discontinuation due to drug-related adverse events, frequency of drug-related events, number of breakthrough fungal infections, and number of successfully treated baseline fungal infections in patients treated with these regimens.
* Compare incidence of required dose increase due to inadequate clinical response in patients treated with these regimens.
* Compare the time to resolution of fever in patients treated with these regimens.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to high-risk (prior allogeneic bone marrow transplantation or prior chemotherapy for relapse of acute leukemia) vs low-risk and prior prophylactic antifungal therapy during chemotherapy (yes vs no). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive caspofungin acetate IV over 1 hour followed by placebo IV over 2 hours.
* Arm II: Patients receive placebo IV over 1 hour followed by amphotericin B liposomal IV over 2 hours.

Treatment repeats daily for up to 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed at 7 and 14 days after study drug discontinuation.

PROJECTED ACCRUAL: A total of 1060 patients (530 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Leukemia, lymphoma, or other cancer that has been previously treated with chemotherapy or bone marrow or peripheral blood stem cell transplantation
* Absolute neutrophil count less than 500/mm^3 for past 96 hours and not expected to recover in next 48 hours
* Received at least 96 hours of parenteral systemic antibacterial therapy
* Fever greater than 38.0 degrees Celsius
* Adequately managed bacterial infection allowed if all of the following are true:

  * Negative blood cultures
  * Received at least 5 days of antibiotics to which any bacterial isolates are sensitive
  * Surgical drainage of any abscess fluid or surgical debridement of infected tissues
  * Removal of infected catheters
* No invasive fungal infection
* Not previously enrolled on this study

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Performance status:

* Karnofsky 30-100%

Life expectancy:

* At least 5 days

Hematopoietic:

* Platelet count at least 5,000/mm^3
* INR no greater than 1.6 (no greater than 4.0 if receiving anticoagulants)

Hepatic:

* Bilirubin no greater than 3 times upper limit of normal (ULN)
* AST or ALT no greater than 5 times ULN
* Alkaline phosphatase no greater than 3 times ULN
* No acute hepatitis or cirrhosis

Renal:

* Not specified

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception
* No allergy, hypersensitivity, or prior serious reaction to any echinocandin antifungal or amphotericin B formulation
* No other condition or illness that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* See Disease Characteristics
* No concurrent investigational antineoplastic therapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* At least 10 days since prior parenteral amphotericin B
* At least 14 days since prior investigational antibiotic, antifungal, or immunosuppressive drug
* No concurrent rifampin or cyclosporine
* No other concurrent investigational antibiotic, antifungal, or immunosuppressive drug
* No concurrent alcohol

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-08; Primary Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kent Sepkowitz, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Walsh TJ, Teppler H, Donowitz GR, Maertens JA, Baden LR, Dmoszynska A, Cornely OA, Bourque MR, Lupinacci RJ, Sable CA, dePauw BE. Caspofungin versus liposomal amphotericin B for empirical antifungal therapy in patients with persistent fever and neutropenia. N Engl J Med. 2004 Sep 30;351(14):1391-402. doi: 10.1056/NEJMoa040446. PMID 15459300